CLINICAL TRIAL: NCT01863823
Title: Director of Research Division
Brief Title: The Effective Treatment of Oral Helicobacter Pylori With the Success Rate of Gastric Eradication
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ameritek USA (Industry)
Responsible Party: Principal Investigator, K C Yee, Director of Research Division, Ameritek USA
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: AmeritekUsa; Ameritek USA (Registry Identifier: Ameritek USA)
Record Dates: First submitted 2013-05-10; First posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Oral Helicobacter Pylori
Keywords: Symptomatic patients; asymptomatic individuals; clinical trial
MeSH Terms: interventions — Amoxicillin; Tetracyclines

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amoxicillin and Tetracyclines (Other): drug treatment
  Interventions: Drug: Amoxicillin and Tetracyclines
- Mouth washing (Other): Mouth washing
  Interventions: Drug: Mouth washing

INTERVENTIONS:
Drug: Amoxicillin and Tetracyclines — 202 symptomatic and 148 asymptomatic individuals were recruited and tested using Saliva H. pylori antigen tests (HPS), H. pylori flagellin (HPF), the urea breathe test (UBT) and the polymerase chain reaction (PCR) test. Test subjects also received various treatments.
  Other Names: dBest
  Arms: Amoxicillin and Tetracyclines
Drug: Mouth washing — Two time washing mouth per day
  Other Names: dBest
  Arms: Mouth washing

SUMMARY:
1. Gastric eradication has no effective on oral H. pylori infection.
2. Treatment of oral infection increase success rate of eradication on stomach infection.

DETAILED DESCRIPTION:
Objective: The present study was aimed to explore the relationship of Helicobacter pylori(H. pylori) of the oral cavity with the success rate eradication of gastric H. pylori infection.

Study Design and Setting: 202 symptomatic and 148 asymptomatic individuals were recruited and tested using Saliva H. pylori antigen tests (HPS), H. pylori flagellin (HPF), the urea breathe test (UBT) and the polymerase chain reaction (PCR) test. Test subjects also received various treatments.

We collected data of HPS, HPF , PCR and UBT before treatment on 202 symptomatic patients and 148 asymptomatic individual groups. After drug treatment, we run HPS, HPF, PCR and UBT tests. If the tests of HPS, HPF and PCR show negative that indicate success of oral H.pylori eradication. If the test of UBT show negative that indicate success of stomach H.pyloi eradication. We also compare the suceess rate of eradication on stomach infection with and without oral H. pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* patients with gastrointestinal complaints

Exclusion Criteria:

* patients who had taken any antibiotics and/or proton pump inhibitors within four weeks prior to sample collection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Success Rate | 12 months

SECONDARY OUTCOMES:
Diagnostic | 6 months

OTHER OUTCOMES:
Agreement of diagnostic and success rate of gastric eradication | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing University First Hospital, Beijiang, China

REFERENCES:
- [Derived] Wang XM, Yee KC, Hazeki-Taylor N, Li J, Fu HY, Huang ML, Zhang GY. Oral Helicobacter pylori, its relationship to successful eradication of gastric H. pylori and saliva culture confirmation. J Physiol Pharmacol. 2014 Aug;65(4):559-66. PMID 25179088